CLINICAL TRIAL: NCT01581450
Title: Evaluation of Antihyperalgesic and Analgesic Effects of 35% Nitrous Oxide in a Human Model of Electrically Evoked Hyperalgesia and Pain
Brief Title: Hyperalgesia and Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: ORION Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-000966-37
Record Dates: First submitted 2011-11-30; First posted 2012-04-20 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hyperalgesia
Keywords: Hyperalgesia and pain
MeSH Terms: conditions — Hyperalgesia; Pain | interventions — Nitrous Oxide; kalinox

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tested drug (Experimental): Remifentanil at 0.1 µg/kg/min Tested drug (N2O 35%): 35%/15%/50% N2O/N2/O2
  Interventions: Drug: Nitrous Oxide
- Gas Active control (Active Comparator): Remifentanil at 0.1 µg/kg/min Gas active control (N2O 50%):50%/50% N2O/O2
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — 35%
  Arms: Tested drug
Drug: Nitrous Oxide — 50%
  Other Names: Kalinox
  Arms: Gas Active control

SUMMARY:
Evaluation of the effects of 35%/15%/50% N2O/N2/O2 mixtures on the area of hyperalgesia induced by remifentanil in the CCES (Continuous Cutaneous Electrical Stimulation) model in 20 healthy volunteers.

The duration of participation for each volunteer is expected to be around 9 weeks with the performance of 4 experimental session 2 weeks apart.

The selection visit will last half a day; each experimental session will last half a day; the study end will last 2 hours maximum.

DETAILED DESCRIPTION:
Single site, exploratory, comparative, double-blind, randomised, cross-over study. Three physicians will be involved in the conduct of this study:

* Physician 1 will include and randomise the subjects, prepare and administer the study products (namely Investigational Medicinal Products (IMPs)) in an open manner and will assess subject safety.
* Physician 2, kept IMP blinded, will perform all evaluation measurements and sedation assessments during all experimental sessions. Physician 2 will always be the same person throughout the whole study period.
* Physician 3 will be available if needed to reinforce subject safety

Design: A group of 20 assessable subjects who will undergo 4 randomised experimental sessions of CCES on 4 separate study days, 2 weeks apart preceded by a 2 week period between selection and first experimental session and followed by a 1 week period between last experimental session and study end.

After the selection visit, each visit corresponds to one of the 4 experimental sessions named A, B, C, D differing by the gas mixture inhaled and the intravenous medicine administered.

The order of these experimental sessions A, B, C, D, will be assigned according to a pre-established list that the investigator will not know.

Each experimental session includes a set-up-phase followed by an evaluation phase.

The set up phase will last 20 mn during each an electrical stimulation will generate a spontaneous pain: every 2 minutes the electrical stimulation will increase and the subject will be asked to rate the pain on a visual scale from 0 to 100. When a stable levels of pain intensity will be reached, the regimen of the electrical stimulation will be kept constant up to the end of the experimental session.

The Evaluation phase will last 160 mn : the electrical stimulation will be constant during 160 mn as detailed above. During this phase the subject will inhale a gas mixture with a face mask during 60 minutes combined with an intravenous administration of medicine during 30 mn starting at the same time.

Every 5 minutes the subject will be asked to rate the pain and at predefined times the spontaneous pain and the area of allodynia and hyperalgesia will be measured and recorded as well as safety parameters (transcutaneous oxygen saturation, respiratory parameters, sedation score, blood pressure and heart rate).

The 4 experimental sessions named A, B, C, D differ by the gas mixture inhaled and the intravenous medicine administered.

For the placebo session, inhaled gas mixture will be 50%/50% N2/O2 and intravenous administration will be an isotonic saline solution.

For the three other sessions, inhaled gas mixture will differ from a session to the other one (35%/15%/50% N2O/N2/O2 or 50%/50% N2/O2 or 50%/50% N2O/O2), and remifentanil will be administered intravenously at each of these sessions.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian healthy male
* Able to feel a distinct pin-pick sensation on normal skin
* Subject willing and able to complete the requirements of this study
* Written informed consent signed prior to any study related procedures

Exclusion Criteria:

* History of any past or current renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine haematological, neurological, psychiatric disease or other disorders
* Any significant history of allergic disease
* Acute skin disease, lesions, acute sunburn, extensive tattoos or scars
* Donation of blood within the previous 3 months
* participation in any other clinical study within the previous 4 weeks.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Hyperalgesia | at T0, T10, T25, T40, T55, T70, T95, T110, T125, T140 and T155 minutes at each experimental session which will last half day
  - Hyperalgesia will be assessed by using a metal rod,(in unit cm).

SECONDARY OUTCOMES:
transcutaneous oxygen saturation | From T0 to T160 minutes, at 5 minute intervals at each experimental session which will last half day
  By monitoring pulse oximetry device
respiration rate | From T0 to T160 minutes, at 5 minute intervals at each experimental session which will last half day
  Respiration rate
systolic and diastolic blood pressures | From T0 to T160 minutes, at 5 minute intervals at each experimental session which will last half day
  systolic and diastolic blood pressures
Heart rate | From T0 to T160 minutes, at 5 minute intervals at each experimental session which will last half day
  Measured by cardioscope
sedation score | From T0 to T160 minutes, at 5 minute intervals at each experimental session which will last half day
  sedation score

CONTACTS AND LOCATIONS:
Overall Officials: Andreas WEHRFRITZ, MD, Principal Investigator — University of Erlangen-Nürnberg, Germany
Locations (1):
- University of Erlangen - Nürnberg, Erlangen, Germany

REFERENCES:
- [Result] Wehrfritz A, Bauer M, Noel N, Ramirez-Gil JF, Ihmsen H, Prottengeier J, Schuttler J, Bessiere B. Evaluation of antihyperalgesic and analgesic effects of 35% nitrous oxide when combined with remifentanil: A randomised phase 1 trial in volunteers. Eur J Anaesthesiol. 2021 Dec 1;38(12):1230-1241. doi: 10.1097/EJA.0000000000001468. PMID 34735395